CLINICAL TRIAL: NCT07100717
Title: Compassion Fatigue and Compassion Satisfaction Among Nurses in Oman: Intervention Study
Brief Title: Intervention Study on Compassion Fatigue and Satisfaction in Omani Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oman Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: MoH/CSR/25/29865
Record Dates: First submitted 2025-07-16; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Registered Nurses; Compassion Fatigue; Occupational Stress; Mental Health
Keywords: Nurses; Oman; Compassion Fatigue; Compassion Satisfaction; Burnout; Intervention; Healthcare Workers; Mental Health
MeSH Terms: conditions — Compassion Fatigue; Occupational Stress; Psychological Well-Being; Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mindfulness-based self-care (MBSC) program (Other): A 2-day workshop and self-mindfulness practices
  Interventions: Behavioral: 2-days workshop and self-mindfulness practices

INTERVENTIONS:
Behavioral: 2-days workshop and self-mindfulness practices — Participants will attend 2-days face-to-face workshop on mindfulness-based self-care (MBSC) program. After the completion of the 2-days workshop, the participants will be required to complete self-mindfulness practices within a period of 4 weeks

SUMMARY:
The purpose of this study is to assess the level of compassion fatigue and compassion satisfaction among nurses working at Ministry of Health hospitals. It will also examine the significant demographics, work-related contributing factors, and the impact of a mindfulness self-care program on nurses' compassion fatigue and compassion satisfaction level.

DETAILED DESCRIPTION:
A cross-sectional design will be used for the first stage of the study. A pre-post- intervention study will be utilized for the second stage of the study. A convenience sample of 361 nurses from six governmental hospitals of the Ministry of Health will be enrolled for the first stage of the study. A minimum of (50) participants, from the hospital with the highest level of compassion fatigue will be included in the intervention stage of the study. An integrated guided mindfulness intervention will be implemented, which will include a 2-day face-to-face workshop and self-practice activities.

The Professional Quality of Life (ProQOL), version 5 (Stamm, 2010), which measures compassion fatigue, will be used in addition to the participants demographic and work-related contributing factors.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses (males & females; Omani & Non-Omani)
* With direct patient care
* A minimum of six months experience in same hospital's unit/word
* Currently not receiving psychiatric or mental therapy

Exclusion Criteria:

* Registered nurses with no direct patient care
* Less than six months of work experience in a hospital unit/word
* Currently under psychiatric or mental therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-21 (Estimated); Primary Completion 2026-01-29 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Compassion Fatigue | From enrollment to the end of Mindfulness-self practices at 4 weeks
  The compassion fatigue level will be measured using The Professional Quality of Life (ProQOL) scale, version 5. The ProQOL is a 5-point Likert well-known scale (1= never, 5= very often) that utilized globally to assess the compassion fatigue (Babaei & Haratian, 2020; Hooper et al., 2010). The instrument consists of three subscales, which are compassion satisfaction, burnout, and secondary traumatic stress. The scale is constructed of 30-items; where 10 items measuring each subscale (i.e. compassion satisfaction, burnout, and secondary traumatic stress). The response of instruments' items are based on the respondent's opinions and feelings for the last 30 days (Babaei & Haratian, 2020). The cut-scores are set around the 25th and 75th percentiles. The instrument demonstrated a good construct validity as well as good internal consistency of reliability for each subscale with Cronbach alphas of 0.87, 0.72, and 0.80, respectively (Hooper et al., 2010).
Compassion Satisfaction | From enrollment to the end of mindfulness-self practice sessions at 4 weeks
  Compassion satisfaction level will be measured by The Professional Quality of Life (ProQOL) scale, version 5. The instrument consists of three subscales, which are compassion satisfaction, burnout, and secondary traumatic stress. The response of instruments' items are based on the respondent's opinions and feelings for the last 30 days (Babaei & Haratian, 2020). The cut-scores are set around the 25th and 75th percentiles. The instrument demonstrated a good construct validity as well as good internal consistency of reliability for each subscale with Cronbach alphas of 0.87, 0.72, and 0.80, respectively (Hooper et al., 2010).

SECONDARY OUTCOMES:
Demographic and work-related characteristics | At the end of mindfulness-self practice at 4 weeks
  The demographic and work-related characteristics will be assessed using a developed questionnaire for the purpose of this study. The questionnaire includes items of age, gender, marital status, education degree, years of experience, and working department/word/unit.

CONTACTS AND LOCATIONS:
Overall Officials: Shawana M Al Harrasi, PhD, Principal Investigator — Oman College of Health Sciences
Locations (1):
- MoH Regional Hospital, Rustaq, South Batinah, Oman

IPD SHARING:
Plan to Share IPD: No